CLINICAL TRIAL: NCT03228147
Title: Sensory Evaluation of a New Oral Nutrition Supplement in Patients at Risk for Mucositis
Brief Title: Sensory Evaluation of Oral Nutrition Supplements in Patients at Risk for Mucositis Undergoing Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 071701; NCI-2017-01151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20170000485; 071701 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2017-07-18; First posted 2017-07-24 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Esophagitis; Malignant Neoplasm; Mucositis
MeSH Terms: conditions — Esophagitis; Neoplasms; Mucositis | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (nutrition supplement) (Experimental): Patients receive 10 different nutrition supplements PO and complete questionnaires based on each sample in a single session over 60-90 minutes.
  Interventions: Dietary Supplement: Nutritional Supplementation; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Nutritional Supplementation — Given PO
  Other Names: Supplementation
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies sensory evaluation of oral nutrition supplements in patients at risk for mucositis undergoing cancer treatment. Sensory evaluation may help to obtain input about new oral nutritional supplements that may increase nutrient intake and maintain or improve nutritional status, functional capacity, and quality of life in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify two products (one from the creamy shake category and one from the tea category) with the highest total average score that will be selected to move onto further testing.

OUTLINE:

Patients receive 10 different nutrition supplements orally (PO) and complete questionnaires based on each sample in a single session over 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cancer treatment (chemotherapy, radiotherapy, and/or immunotherapy)
* At risk for mucositis OR with stage I mucositis or esophagitis (i.e. radiotherapy to the head, neck, esophagus or lung OR treatment with fluorouracil (5-FU) or other chemotherapeutic agents that are known to cause mucositis or esophagitis) or at risk for xerostomia
* Within the first 3 weeks of initiation of a new type of therapy
* Able to read and write in English
* Able to provide written informed consent

Exclusion Criteria:

* Food allergy to any component of the supplement
* Inability to taste or smell due to medication or health condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
A creamy shake product with the highest total average nutrition supplement scores as assessed by questionnaires | Up to 1 year
  Will identify one product from the creamy shake category with the highest total average score that will be selected to move onto further testing. The subjective assessments of each formula will be assessed and mean, standard deviation and range will be calculated for each response. There will be subjective evaluation of acceptance of the overall sensory attributes and flavor liking (9-point scale), open-ended description of sensory attributes and effects (aroma, flavor, aftertaste, off-flavors), flavor intensity, sweetness (too little, just about right, too thick) 5-point scale. In-mouth sensations (cooling, tingling, mouth wetting, refreshing, soothing, wetting) 9-point scale.
A tea product with the highest total average nutrition supplement scores as assessed by questionnaires | Up to 1 year
  Will identify one product from the tea category with the highest total average score that will be selected to move onto further testing. The subjective assessments of each formula will be assessed and mean, standard deviation and range will be calculated for each response. There will be subjective evaluation of acceptance of the overall sensory attributes and flavor liking (9-point scale), open-ended description of sensory attributes and effects (aroma, flavor, aftertaste, off-flavors), flavor intensity, sweetness (too little, just about right, too thick) 5-point scale. In-mouth sensations (Cooling, tingling, mouth wetting, refreshing, soothing, wetting) 9-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Salma Jabbour, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States